CLINICAL TRIAL: NCT03020225
Title: Protein Bioavailability of Wolffia Globosa (Mankai); Acute Test Meal Effects
Acronym: Mankai
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ben-Gurion University of the Negev (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); University of Leipzig (Other)
Responsible Party: Principal Investigator, Iris Shai, Principle investigator, Ben-Gurion University of the Negev
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BenGurionU
Record Dates: First submitted 2017-01-09; First posted 2017-01-13 (Estimated); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-01

CONDITIONS: Men With Mild Abdominal Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- White cheese (Active Comparator): Reference group- animal protein food source: White cheese (contains 30g protein), intact, plus 250ml mineral water
  Interventions: Dietary Supplement: White cheese
- Green peas (Experimental): Plant food source: Green peas (contains 30g protein), intact, cooked, plus 250ml mineral water
  Interventions: Dietary Supplement: Green peas
- Mankai (Experimental): Plant food source: Wolffia globosa (Mankai, contains 30g protein), intact, cooked, plus 250ml mineral water
  Interventions: Dietary Supplement: Mankai

INTERVENTIONS:
Dietary Supplement: White cheese — animal protein food source: White cheese (contains 30g protein), intact, plus 250ml mineral water
  Arms: White cheese
Dietary Supplement: Green peas — Green peas (contains 30g protein), intact, cooked, plus 250ml mineral water
  Arms: Green peas
Dietary Supplement: Mankai — Wolffia globosa (Mankai, contains 30g protein), intact, cooked, plus 250ml mineral water
  Arms: Mankai

SUMMARY:
The investigators aim to test the protein bioavailability of new specific developed strain of duckweed [Wolffia globose, Mankai] , an aquatic plant, which might serve as a protein source and contains all the 9 essential and the 6 conditional amino acids. The investigators will randomize 36 participants to consume equivalent protein (30gr) content of 3 whole foods items: 1. White cheese (animal protein source, as a reference); 2. Green peas, intact, cooked (plant protein source); 3. Wolffia globosa (Mankai), intact, cooked (plant protein source). The foods will be consumed in the morning, following 12h fasting. The foods will be provided with 250ml mineral water and the blood follow-up frame will be for 3 hours. Primary outcome: Blood amino acid profile.

DETAILED DESCRIPTION:
The investigators aim to test the protein bioavailability of new specific developed strain of duckweed [Wolffia globose, Mankai], an aquatic plant, which might serve as a protein source and contains all the 9 essential and the 6 conditional amino acids. "Mankai" [(Generally recognized as safe (GRAS)] is a cultivated strain of Wolffia globosa, which is an aquatic plant, part of the family of plants known commonly as duckweeds. Duckweeds are very simple flowering aquatic plants which float on or just beneath the surface of still or slow-moving bodies of water. There is a long history of the use of Wolffia species, in particular Wolffia Globosa, as food, especially in Southeast Asia: Burma, Laos and northern Thailand, where it has been used as a vegetable for many generations. There are numerous ways of W. globosa consumption and a variety of recipes, using it either as a main ingredient (such as Wolffia crisps or "kaeng pum" - a popular vegetable dish in northeastern Thailand) or incorporating it in other foods (e.g. Wolffia-meat ball, fermented Wolffia-meat sausage, Wolffia rice noodle, Wolffia cookies, Wolffia bread, and various soups and salads). Along with its long history as a food source in Southeast Asia, it is recognized as an edible vegetable for humans in several databases, including the United States Department of Agriculture (USDA 2014) GRIN database and a database dedicated to tropical species. The nutritional composition of Mankai has been determined and found to be high in protein, containing all the essential and conditionally essential amino acids, dietary fibers and several vitamins and minerals. In a recent safety study, which aimed to test the safety of Mankai administration within and 3 times of the amount approved in the GRAS, 4 groups of female SD rats were orally administered for 4 consecutive days a daily dose of Mankai at three dose levels of 1700, 2500 and 3400mg/kg of Mankai, equivalent to 20, 40 and 60 gr/day human dose, respectively. Clinical (e.g body weight, food intake, morbidity/mortality, toxic signs), pathological (post mortem gross pathology examination) and long list of blood biochemical indicators (e.g liver status biomarkers, stress indicators, minerals) did not show any adverse effects. The results indicate that repeated four day Mankai administration did not cause adverse effects. Unexpectedly, high doses even suggested beneficial results with anti-glycemic effects. Mankai was found to have a high digestibility profile (89%) according to Protein digestibility-corrected amino acid score (PDCAAS) Eurofins tests. However, its human nutrient bioavailability has not been examined yet. For the proposed test, Mankai (grown by Hinoman Ltd., Israel) will be provided as a fresh, whole, product.

Methods: 36 men will be randomized to consume the following food items, which will be equivalent to 30gr protein, after 12h night fasting:

1. Reference group: animal protein food source: White cheese, intact, plus 250ml mineral water
2. Test group 1: plant food source: Green peas, intact, cooked, plus 250ml mineral water
3. Test group 2: plant food source: Wolffia globosa (Mankai), intact, cooked, plus 250ml mineral water

The participants will be asked to maintain a stable diet (according to guidelines that will be provided) for 3 days prior to the test meal. Blood samples will be taken at times 0, 30, 90, and 180 minutes.

ELIGIBILITY:
Inclusion Criteria:

* age >30 years; abdominal adiposity (waist circumference: men > 102 cm, women > 88 cm) or dyslipidemia

Exclusion Criteria:

* triglycerides>400 mg/dL; serum creatinine>2 mg/dL;
* disturbed liver function;
* pregnant or lactating women;
* presence of active cancer, is receiving or received chemotherapy in the last three years; participation in another trial;
* participants who are treated with Coumadin (warfarin)

Min Age: 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-12; Primary Completion 2017-02 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shai, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- nuclear research center Negev, Dimona, Israel

REFERENCES:
- [Derived] Kaplan A, Zelicha H, Tsaban G, Yaskolka Meir A, Rinott E, Kovsan J, Novack L, Thiery J, Ceglarek U, Burkhardt R, Willenberg A, Tirosh A, Cabantchik I, Stampfer MJ, Shai I. Protein bioavailability of Wolffia globosa duckweed, a novel aquatic plant - A randomized controlled trial. Clin Nutr. 2019 Dec;38(6):2576-2582. doi: 10.1016/j.clnu.2018.12.009. Epub 2018 Dec 11. PMID 30591380

RESULTS

PARTICIPANT FLOW:
Recruitment Details: https://www.ncbi.nlm.nih.gov/pubmed/30591380
Pre-assignment Details: https://www.ncbi.nlm.nih.gov/pubmed/30591380
Period: Overall Study
Arm/Group | White Cheese | Green Peas | Mankai
Started | 12 | 11 | 13
Completed | 12 | 11 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: https://www.ncbi.nlm.nih.gov/pubmed/30591380
Groups:
- Total: Total of all reporting groups
Arm/Group | White Cheese | Green Peas | Mankai | Total
Number analyzed (Participants) | 12 | 11 | 13 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (8.8) | 49.5 (12.1) | 48.9 (11) | 48.8 (10.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  number of man (%) | 12 | 11 | 13 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Israel | 12 | 11 | 13 | 36
Histidine (EAA) [Mean (Standard Deviation); unit: µmol/L] | 31.1 (4.1) | 31.3 (4.1) | 30 (2.9) | 30.7 (3.7)
Tryptophan (EAA) [Mean (Standard Deviation); unit: µmol/L] | 14.2 (2.9) | 13.8 (3.5) | 12.4 (2.5) | 13.4 (3)
Phenylalanine (EAA) [Mean (Standard Deviation); unit: µmol/L] | 67.4 (13.5) | 60.3 (10.2) | 63.4 (8.5) | 63.8 (10.9)
Methionine (EAA) [Mean (Standard Deviation); unit: µmol/L] | 30.3 (7.4) | 25.6 (4.2) | 28.2 (6.1) | 28.1 (6.2)
Threonine (EAA) [Mean (Standard Deviation); unit: µmol/L] | 31.2 (6.7) | 29.9 (6.8) | 30.2 (5.7) | 30.5 (6.2)
Lysine (EAA) [Mean (Standard Deviation); unit: µmol/L] | 81 (24.9) | 73.2 (22.2) | 72.7 (19.5) | 75.6 (21.9)
Valine (EAA) [Mean (Standard Deviation); unit: µmol/L] | 187.1 (31.2) | 179.3 (36.3) | 184.4 (25) | 183.7 (30.2)
Isoleucine/leucine (EAA) [Mean (Standard Deviation); unit: µmol/L] | 141.8 (27.2) | 129 (26.6) | 139.7 (19.6) | 137.1 (24.5)

OUTCOME MEASURES:

1. Primary Outcome: Amino Acid Profile (Blood Biomarkers)
Description: will be analysed by metabolomic for amino acid profile (trajectory)
Time Frame: 3 hours
Population: Essential amino acids (mmol/L) for the 3 groups
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- White Cheese: Essential amino acids (mmol/L)
- Green Peas; Mankai: Essential amino acids
Arm/Group | White Cheese | Green Peas | Mankai
Number analyzed (Participants) | 12 | 11 | 13
mmol/L | 31.1 (4.1) | 31.1 (4.1) | 30 (2.9)

2. Secondary Outcome: Glycemic Profile
Description: glucose (blood biomarkers)
Time Frame: 3 hours
Population: glucose
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- White Cheese; Green Peas; Mankai: blood biomarkers of glycemia
Arm/Group | White Cheese | Green Peas | Mankai
Number analyzed (Participants) | 12 | 11 | 13
mg/dL | 97.5 (13.4) | 96 (9.2) | 96.7 (9.4)

3. Secondary Outcome: Lipid Profile
Description: HDL cholesterol fractions (blood biomarkers)
Time Frame: 3 hours
Population: cholesterol fractions
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- White Cheese; Green Peas; Mankai: cholesterol fractions
Arm/Group | White Cheese | Green Peas | Mankai
Number analyzed (Participants) | 12 | 11 | 13
mg/dL | 45.3 (9.9) | 41.9 (9.3) | 44.4 (7.8)

4. Secondary Outcome: Liver Function
Description: ALT (blood biomarkers)
Time Frame: 3 hours
Population: ALT
Measure: Mean (Standard Deviation); unit: U/l
Groups:
- Soft Cheese; Green Peas; Mankai: ALT measured in blood
Arm/Group | Soft Cheese | Green Peas | Mankai
Number analyzed (Participants) | 12 | 11 | 13
U/l | 43.2 (13.2) | 42.3 (21.1) | 46 (19.5)

5. Secondary Outcome: Minerals
Description: potassium (blood measures)
Time Frame: 3 hours
Population: potassium
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- White Cheese; Green Peas; Mankai: potassium levels
Arm/Group | White Cheese | Green Peas | Mankai
Number analyzed (Participants) | 12 | 11 | 13
mmol/L | 4.5 (0.2) | 4.7 (0.3) | 4.5 (0.2)

6. Secondary Outcome: Vitamins
Description: B12 (blood measures)
Time Frame: 3 hours
Population: B12
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- White Cheese; Green Peas; Mankai: Vitamin B12 (blood measures)
Arm/Group | White Cheese | Green Peas | Mankai
Number analyzed (Participants) | 12 | 11 | 13
pg/mL | 371.1 (146.4) | 473 (144.1) | 423 (220.4)

7. Secondary Outcome: Glycemic Profile-Insulin
Description: Insulin (blood biomarker)
Time Frame: 3 hours
Population: Insulin
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | White Cheese | Green Peas | Mankai
Number analyzed (Participants) | 12 | 11 | 13
mg/dL | 97.5 (13.4) | 96 (9.2) | 96.7 (9.4)

8. Secondary Outcome: Triglycerides
Description: Triglycerides levels- Lipid profile
Time Frame: 3 hours
Population: Triglycerides
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- White Cheese; Green Peas; Mankai: Triglycerides
Arm/Group | White Cheese | Green Peas | Mankai
Number analyzed (Participants) | 12 | 11 | 13
mg/dl | 172.2 (77) | 198 (111.7) | 207.9 (83)

9. Secondary Outcome: Liver Enzymes- ASAT
Description: ASAT - Liver enzymes
Time Frame: 3 hours
Population: ASAT
Measure: Mean (Standard Deviation); unit: μKat/L
Groups:
- Soft Cheese; Green Peas: ASATmeasured in blood
- Mankai: ASAT measured in blood
Arm/Group | Soft Cheese | Green Peas | Mankai
Number analyzed (Participants) | 12 | 11 | 13
μKat/L | 0.53 (0.09) | 0.49 (0.09) | 0.51 (0.18)

10. Secondary Outcome: Magnesium
Description: Magnesium levels
Time Frame: 3 hours
Population: Magnesium levels
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- White Cheese; Green Peas; Mankai: Magnesium levels
Arm/Group | White Cheese | Green Peas | Mankai
Number analyzed (Participants) | 12 | 11 | 13
mmol/L | 0.87 (0.072) | 0.95 (0.28) | 0.91 (0.054)

ADVERSE EVENTS:
Time Frame: 3 hours
Arm/Group | White Cheese | Green Peas | Mankai
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT03020225/Prot_SAP_000.pdf